CLINICAL TRIAL: NCT00633477
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of TAK-242 Versus Placebo in Subjects With Sepsis-Induced Cardiovascular and Respiratory Failure
Brief Title: Efficacy and Safety of Resatorvid in Patients With Sepsis-induced Cardiovascular and Respiratory Failure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision; No Safety Or Efficacy Concerns.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-242_301; 2007-005687-27 (EudraCT Number); U1111-1127-6016 (Registry Identifier: WHO)
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Sepsis
Keywords: Systemic Inflammatory Response Syndrome; Septic Shock; Septicemia; Drug Therapy
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome; Shock, Septic | interventions — ethyl 6-(N-(2-chloro-4-fluorophenyl)sulfamoyl)cyclohex-1-ene-1-carboxylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resatorvid 2.4 mg/kg/day (Experimental)
  Interventions: Drug: Resatorvid
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resatorvid — Resatorvid 1.2 mg/kg emulsion, injection for 30 minutes and resatorvid 2.4 mg/kg per-day emulsion, injection, continuous infusion for 96 hours.
  Other Names: TAK-242
  Arms: Resatorvid 2.4 mg/kg/day
Drug: Placebo — Resatorvid placebo-matching emulsion, injection for 30 minutes and resatorvid placebo-matching emulsion, injection, continuous infusion for 96 hours.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of resatorvid on subjects with sepsis.

DETAILED DESCRIPTION:
Sepsis is a major cause of in-hospital death, with a higher mortality rate than events such as stroke and acute myocardial infarction, each with less than a 20% risk of death in the first 30 days. Sepsis is a clinical condition caused by the innate inflammatory host response to systemic infection that can result in organ failure and potentially death. Under certain circumstances, many components of the innate immune response that are normally involved with host defense can cause cell and tissue damage and subsequently multiple organ failure, the clinical hallmark of severe sepsis.

The host response to infection is characterized by the synthesis and release of proinflammatory cytokines. Cytokines are released by signals transmitted from the surface of inflammatory cells, after binding of pathogen-associated molecules to cell surface pattern recognition receptors known as toll-like receptors.

TAK-242 (resatorvid) is a toll-like receptor 4 inhibitor under clinical development for the treatment of patients with severe sepsis. Study participation is anticipated to be about 28 days, with an additional 9 month follow-up period.

ELIGIBILITY:
Inclusion Criteria

* Suspected or proven bacterial or fungal infection for which patient is receiving parenteral antimicrobial therapy.
* Developed at least 3 of the 4 following systemic inflammatory response syndrome criteria within 36 hours prior to start of study drug administration:

  * A temperature from any site greater than 38°C (greater than 100.4°F) or a core temperature less than 36°C (less than 96.8°F).
  * Heart rate of greater than 90 beats per minute. If subject has a known medical condition (eg, heart block) or is receiving treatment (eg, beta blocker) that would prevent tachycardia, only 2 of the remaining 3 criteria for systemic inflammatory response syndrome must be met.
  * Respiratory rate of greater than 20 breaths per min or arterial partial pressure of carbon dioxide of less than 32 mm Hg or mechanical ventilation for an acute process.
  * A total white blood cell absolute count greater than 12,000 cells per mm3 or less than 4,000 cells/mm3; or a white blood cell differential count showing greater than 10% immature (band) forms.
* Has septic shock diagnosed within 36 hours prior to study drug administration..
* Has developed respiratory failure within 36 hours prior to study drug administration.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria

* Received any investigational compound within 30 days (or 5 half-lives of the drug, whichever is longer) prior to the initiation of the study drug infusion or is participating in another investigational study, not including investigational compound, without prior approval from the Vanderbilt Coordinating Center or the sponsor.
* Currently receiving any immunosuppressive therapy (excluding glucocorticoids) such as methotrexate, azathioprine, anti tumor necrosis factor alpha, or a cancer related chemotherapeutic agent.
* Known history of glucose-6-phosphate dehydrogenase deficiency.
* Methemoglobin level of greater than or equal to 5% at pretreatment period or has a known history of methemoglobinemia.
* Moribund and death is considered imminent.
* Prior to the onset of sepsis, the subject would not otherwise have been expected to survive 28 days or to complete a functional recovery due to a pre-existing unstable medical condition (eg, a recent acute cerebral hemorrhage or infarct, a recent acute unstable myocardial infarction, severe traumatic injury).
* Poorly controlled or metastatic neoplasm.
* The participant, the participant's family or physician is not committed to full aggressive management or the presence of an unstable medical condition makes the receipt of full aggressive management support unlikely in the view of the coordinating center.
* Severe end stage chronic respiratory failure or lung disease that significantly impairs physical functioning equivalent to that of New York Heart Association functional classification III or IV.
* Documented history of moderate to severe chronic heart failure as defined by New York Heart Association functional classification III or IV.
* Received electrocardioversion for a pulse-less rhythm or chest compressions during their current hospitalization.
* Known to be immunocompromised such as subjects with human immunodeficiency virus and a CD4 count less than 50 mm3, primary immune deficiency or chronic lymphocytic leukemia.
* Chronic end stage hepatic failure or significant sequelae of chronic hepatic failure (eg, esophageal varices, jaundice, chronic ascites) or Child-Pugh hepatic impairment Classification C.
* In a chronic vegetative state or has a similar long-term neurological impairment, where continued aggressive care would be unlikely.
* Acute third degree burns involving more than 30% of body surface area within 120 hours of first qualifying organ failure.
* Known hypersensitivity to sulphonamides.
* Known hypersensitivity to components of resatorvid; for example, is allergic to eggs, egg products, or soybeans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (1):
- Nagasaki, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the sudy at 11 centers in Japan and 1 center in the United States from 26 February 2008 to 20 February 2009 (day the decision was taken to terminate the study) .
Pre-assignment Details: Participants who met 3 of the 4 systemic inflammatory response syndrome (SIRS) criteria and receiving parentaeral antimicrobial therapy for bacterial or fungal infection prior to enrollment and met the key organ failure criteria within 36 hours of planned study drug administration were randomized to receive resatorvid or placebo.
Groups:
- Resatorvid: Resatorvid 1.2 mg/kg given as a 30-minute loading dose followed by 2.4 mg/kg/day given as a continuous infusion for 96 hours.
- Placebo: Placebo given as a 30-minute loading dose followed by a continuous infusion for 96 hours.
Period: Overall Study
Arm/Group | Resatorvid | Placebo
Started | 7 (Seven subjects were randomized, however, one was not treated.) | 11
Randomized But Not Treated | 1 | 0
Prematurely Discontinued Study Drug | 1 | 0
Completed Study Through Day 28 | 4 | 8
Completed | 5 (Include all subjects who could be evaluated for 28-d survival.) | 11 (Include all subjects who could be evaluated for 28-d survival.)
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Randomized but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Resatorvid 2.4 mg/kg/Day: Resatorvid 1.2 mg/kg given as a 30-minute loading dose followed by 2.4 mg/kg/day given as a continuous infusion for 96 hours
- Total: Total of all reporting groups
Arm/Group | Resatorvid 2.4 mg/kg/Day | Placebo | Total
Number analyzed (Participants) | 6 | 11 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 76.7 (5.28) | 77.8 (13.56) | 77.4 (11.14)
Age, Customized [Number; unit: Participants]
  18 - <45 | 0 | 0 | 0
  45 - <60 | 0 | 1 | 1
  60 - <75 | 2 | 3 | 5
  ≥75 | 4 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 6 | 7 | 13
Race [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 10 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
Ethnicity [Number; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 6 | 10 | 16
Weight [Mean (Standard Deviation); unit: kg] | 54.27 (12.9) | 58.24 (17.1) | 56.84 (15.4)
Height [Mean (Standard Deviation); unit: cm] | 158.3 (6.0) | 160.7 (7.4) | 159.9 (6.9)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 21.46 (3.97) | 22.59 (6.12) | 22.19 (5.36)
Smoking Classification [Number; unit: Participant]
  Never smoked | 2 | 4 | 6
  Current smoker | 0 | 3 | 3
  Ex-smoker | 3 | 4 | 7
  Smoking history not available | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: Mortality regardless of cause at Day 28
Time Frame: Day 28
Population: Participants who received study drug.
Measure: Number; unit: Participants
Arm/Group | Resatorvid | Placebo
Number analyzed (Participants) | 6 | 11
Participants
  Number participants Analyzed | 6 | 11
  Number Alive | 4 | 8
  Number not alive | 2 | 3

2. Primary Outcome: All-cause Mortality
Description: Mortality regardless of cause at Day 28
Time Frame: Day 28
Population: Participants who received study drug
Measure: Number; unit: Percent of Participant
Arm/Group | Resatorvid | Placebo
Number analyzed (Participants) | 6 | 11
Percent of Participant
  Percent Alive | 66.7 | 72.7
  Percent Not alive | 33.7 | 27.3

3. Secondary Outcome: ICU Free Days
Description: Number days participant was not in ICU
Time Frame: Day 28
Population: This study was terminated early when 17 subjects had received treatment.
Measure: Number; unit: days
Arm/Group | Resatorvid | Placebo
Number analyzed (Participants) | 6 | 11
days | NA — This study was terminated early when only 17 subjects had received treatment. | NA — This study was terminated early when only 17 subjects had received treatment.

4. Secondary Outcome: Vasopressor Free Days.
Description: Number days participant did not need vasopressors.
Time Frame: Day 28
Population: This study was terminated early when 17 subjects had received treatment.
Measure: Number; unit: days
Arm/Group | Resatorvid | Placebo
Number analyzed (Participants) | 6 | 11
days | NA — This study was terminated early when 17 subjects had received treatment. | NA — This study was terminated early when 17 subjects had received treatment.

5. Secondary Outcome: Ventilator Free Days.
Description: Number days participant was not on Ventilattor support.
Time Frame: Day 28
Population: This study was terminated early when 17 subjects had received treatment.
Measure: Number; unit: Days
Arm/Group | Resatorvid | Placebo
Number analyzed (Participants) | 6 | 11
Days | NA — This study was terminated early when 17 subjects had received treatment. | NA — This study was terminated early when 17 subjects had received treatment.

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Resatorvid | Placebo
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/11
Other Adverse Events (participants affected / at risk) | 4/6 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Resatorvid (N=6) | Placebo (N=11)
Sepsis (Infections and infestations) | 0 | 2 — Death??
Septic shcok (Infections and infestations) | 1 | 0
Anoxic encephalopathy (Nervous system disorders) | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Renal failure Acute (Renal and urinary disorders) | 0 | 1
Inflamation (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Resatorvid (N=6) | Placebo (N=11)
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Atrial Fibrilation (Cardiac disorders) | 0 | 2
Atrial Flutter (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 1/1
Blood Amylase Increased (Investigations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 1 | 0
Blood Cholesterol Increased (Investigations) | 0 | 1
Blood Methaemoglobin present (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
White Blood cell count increased (Investigations) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Respirotory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Disseminated Intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Hypothermia (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Septic shock (Infections and infestations) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.